CLINICAL TRIAL: NCT04161326
Title: Environmental Health and Myopia Prevention and Control: A Longitudinal Study in China
Brief Title: Environmental Health and Myopia Prevention and Control
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: CCPMOH2016-China-0304
Record Dates: First submitted 2019-11-11; First posted 2019-11-13 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Refractive Errors; Myopia (Disorder)
MeSH Terms: conditions — Refractive Errors; Myopia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Myopia is one of the major causes of low visual acuity during childhood. It is generally more prevalent in urban areas than in rural areas. Current evidence does not address our understanding of the myopia incidence and development and associated risk geographic factors, such as green spaces. Therefore, our study aimed to evaluate the association between geographic factors and myopia base on a population-based large-scaled cohort design.

ELIGIBILITY:
Inclusion Criteria:

* schoolchildren in the 1st to 4th grades

Exclusion Criteria:

* schoolchildren unwilling to participate

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: A prospective longitudinal cohort study of schoolchildren who studied in the 1st to 4th grades was performed.
Sampling Method: Non-Probability Sample
Enrollment: 100000 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
the changes of spherical equivalent refractive (RSE) | up to 3 years
  A multi-linear regression was used.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China